CLINICAL TRIAL: NCT03927937
Title: Tooth Autotransplantation and Bone Dimension Changes. Randomized Clinical Trial.
Brief Title: Tooth Autotransplantation and Bone Dimension Changes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier Rodriguez Lozano, PhD, Universidad de Murcia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/2018
Record Dates: First submitted 2019-04-20; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Bone Loss, Alveolar; Tooth Loss; Bone Atrophy, Alveolar
MeSH Terms: conditions — Alveolar Bone Loss; Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AUTOTRANSPLANTATION TOOTH (Experimental)
  Interventions: Procedure: AUTOTRANSPLANTATION TOOTH

INTERVENTIONS:
Procedure: AUTOTRANSPLANTATION TOOTH — Tooth with imposible prognosis is replace with a healthy tooth from the same patient.

SUMMARY:
Tooth autotransplantation is a treatment option to replace tooth with imposible prognosis. In several cases the receipt site has a reduced bone dimension. This situation may be imposible the treatment with dental implants without bone reconstruction. Autotransplantation seem to improve the anatomic characteristic of the receipt site without any reconstruction approach.

The aim of this study is to evaluate the bone dimension changes followed autotransplantation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Tooth with imposible prognosis
* Plaque index score less than 30%
* No relevant systemic disease
* Smokers (Less than 20 cigars/day)

Exclusion Criteria:

* Pregnancy-Lactation
* Relevant systemic disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in alveolar bone 12 months after tooth autotransplantation | 1 year
  CT-scan evaluation before surgery and 1 year after, measuring the difference in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Murcia, Murcia, Spain